CLINICAL TRIAL: NCT05903365
Title: Etude Observationnelle de Suivi Des Greffes Haplo-identique Dans la Maladie de Fanconi
Brief Title: Observational Follow-up Study of Haplo-identical Transplants in Fanconi Disease
Acronym: HAPLO-FANCONI
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221272
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-04

CONDITIONS: Fanconi Syndrome
MeSH Terms: conditions — Fanconi Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Fanconi disease
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Additional blood samples at J100, M6, M12, M24

SUMMARY:
This observational protocol will allow for an independent, prospective evaluation of the improvement in survival of patients with Fanconi disease in hematological deadlock due to the absence of an HLA-identical donor and having received a haploidentical transplant.

DETAILED DESCRIPTION:
Fanconi's disease is characterised by a constitutional defect in DNA repair which results in the occurrence of bone marrow failure and haematological malignancies, mainly myeloid: at the age of 40, the cumulative incidence of these two types of pathology reaches almost 100%. The only curative treatment for haemtalogocial diseases is allogenic hematopoietic stem cell transplant. Transplantation modalities must be adapted to the particular susceptibility of these patients to DNA bridging agents and radiotherapy. HSC transplantation is indicated with an unaffected matched related or matched unrelated donor when the patient has severe bone marrow failure or a poor prognostic clonal evolution (cytogenetic evolution or proven haemopathy). Alternative transplants (9/10 pheno-identical, haplo-identical and placental blood donors) were no longer proposed in most cases due to the frequency of severe complications (graft-versus-host disease, viral infections) and the catastrophic medium-term survival of around 40% (Dufort, Bone Marrow Transplant 2012, Gluckman Biol Blood Marrow Transplant. 2007). The development over the last decade of new haploidentical or phenoidentical 9/10 transplant protocols with unmodified grafts and GVH prophylaxis with post-transplant cyclosphosphamide or ex vivo T-depletion adapted to the particular susceptibility of patients with Fanconi disease has reduced the incidence of these severe complications.

This observational protocol will allow for an independent, prospective evaluation of the improvement in survival of patients with Fanconi disease in hematological deadlock due to the absence of an HLA-identical donor and having received a haploidentical transplant

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fanconi disease confirmed by chromosome breakage test and/or genetic analysis
* aged between 6 months and 60 years
* with severe pancytopenia (2 of the following criteria: reticulocytes < 60 G/L, PNN < 0.5 G/L and/or platelets < 20 G/L or patients with more than 6 transfusions in the last 12 months)
* with clonal progression (poor prognostic cytogenetics, myelodysplastic syndrome or acute leukaemia)
* with an unaffected haploidentical donor
* having signed the consent after having read the information note, consent of both parents for minors, of the guardian for patients under guardianship
* having a social security scheme (beneficiary or entitled person)

Exclusion Criteria:

* with an unaffected matched related or HLA 10/10 matched unrelated donnor
* under guardianship

Ages: 6 Months to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patient with Fanconi disease
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Overall Survival Rate | 2 years after transplant

SECONDARY OUTCOMES:
Engraftment | At day 100
  Engraftment at least 3 consecutive days with neutrophils > 0.5 G/L and 7 consecutive days with platelets > 20 G/L, with predominantly whole blood donor chimerism
Absolute neutrophils count | At 1 month
Absolute neutrophils count | At 3 months
Absolute neutrophils count | At 6 months
Absolute neutrophils count | At 12 months
Absolute neutrophils count | At 24 months
Absolute number of platelets | At 1 month
Absolute number of platelets | At 3 months
Absolute number of platelets | At 6 months
Absolute number of platelets | At 12 months
Absolute number of platelets | At 24 months
Incidence of grade 2 to 4 Acute Graft versus Host Disease | At 3 months
Incidence of Acute cortico-resistant Graft versus Host Disease | At 3 months
Incidence of Chronic Graft versus Host Disease | At 24 months
Incidence of relapse | At 12 months
Incidence of relapse | At 24 months
Progression free survival | At 12 months
Progression free survival | At 24 months
Incidence of reactivation of cytomegalovirus infection | At 12 months
Incidence of reactivation of Epstein Barr virus infection | At 12 months
Incidence of severe infection of grade 4 and above according to Common Terminology Criteria for Adverse Events (CTCAE) | At 3 months
Incidence of severe infection of grade 4 and above according to Common Terminology Criteria for Adverse Events (CTCAE) | At 6 months
Incidence of severe infection of grade 4 and above according to Common Terminology Criteria for Adverse Events (CTCAE) | At 12 months
Incidence of severe infection of grade 4 and above according to Common Terminology Criteria for Adverse Events (CTCAE) | At 24 months
Graft-versus-host disease-free, relapse-free survival (GRFS) | At 24 months
Incidence of cardiac toxities | At 12 months
Overall survival | At 12 months
Quality of Life questionnaire for adults | At inclusion
  Quality of life will be assessed for adult using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) " EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life questionnaire for adults | At 3 months
  Quality of life will be assessed for adult using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) " EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life questionnaire for adults | At 6 months
  Quality of life will be assessed for adult using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) " EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life questionnaire for adults | At 12 months
  Quality of life will be assessed for adult using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) " EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life questionnaire for adults | At 24 months
  Quality of life will be assessed for adult using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) " EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire for minors | At inclusion
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Quality of life questionnaire for minors | At 3 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Quality of life questionnaire for minors | At 6 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Quality of life questionnaire for minors | At 12 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Quality of life questionnaire for minors | At 24 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning.
Rate of chimerism | At 1 month
Rate of chimerism | At 3 months
Rate of chimerism | At 6 months
Rate of chimerism | At 12 months
Rate of chimerism | At 24 months
Immune reconstitution by analyzing T, B, natural killer (NK), regulatory T cell levels in the peripheral blood | 3 months after transplant
Immune reconstitution by analyzing T, B, natural killer (NK), regulatory T cell levels in the peripheral blood | 6 months after transplant
Immune reconstitution by analyzing T, B, natural killer (NK), regulatory T cell levels in the peripheral blood | 12 months after transplant
Immune reconstitution by analyzing T, B, natural killer (NK), regulatory T cell levels in the peripheral blood | 24 months after transplant
Ferritine levels | At 3 months
Ferritine levels | At 6 months
Ferritine levels | At 12 months
Ferritine levels | At 24 months

IPD SHARING:
Plan to Share IPD: Undecided